CLINICAL TRIAL: NCT03825861
Title: Neoadjuvant FOLFIRINOX in the Treatment of Locally Advanced Gastric Cancer
Acronym: FOLFIRINOX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 933/16
Record Dates: First submitted 2019-01-24; First posted 2019-01-31 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; FOLFIRINOX
MeSH Terms: conditions — Stomach Neoplasms | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOLFIRINOX (Experimental): Oxaliplatin 85mg/m2, Leucovorin 200mg/m2, Irinotecan 180mg/m2, 5-FU 400mg/m2 bolus followed by 2400mg/m2 continuous infusion.
  Interventions: Drug: FOLFIRINOX

INTERVENTIONS:
Drug: FOLFIRINOX — Oxaliplatin 85mg/m2, Leucovorin 200mg/m2, Irinotecan 180mg/m2, 5-FU 400mg/m2 bolus followed by 2400mg/m2 continuous infusion.

SUMMARY:
Phase II single-arm study designed to evaluate the efficacy and safety of preoperative chemotherapy with FOLFIRINOX regimen. The investigators will include 27 patients with resectable locally advanced gastric cancer. They will receive preoperative chemotherapy with FOLFIRINOX regimen by long-term catheter every 14 days for 8 cycles accounting for a total of 4 months of systemic treatment. In the period between 4 and 8 weeks of the last cycle, restaging tests will be performed and if there is no metastatic progression of disease, the patient will undergo surgical treatment with curative intention. The objective is to evaluate whether preoperative treatment with FOLFIRINOX regimen involving continuous infusion and bolus infusion of 5-fluoruracil, irinotecan bolus and oxaliplatin bolus is effective and safe in the neoadjuvant treatment of locally advanced gastric cancer.

The planned recruitment period is 48 months (4 years). There will be a total of 4 months of preoperative chemotherapy. In case of limiting toxicity or disease progression, chemotherapy will be suspended and patients may undergo resection of the primary neoplasia at the discretion of the surgical team of the institution. Patients will be followed for 5 years after entry of the last participant in the protocol for OS and PFS evaluation. The end of the study will occur when the last participant completes their last follow-up visit, which should occur no later than 60 months after enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of gastric adenocarcinoma that is amenable to surgical resection at diagnosis, with locally advanced disease criteria for clinical evaluation (T3 tumors, T4 tumors and / or regional lymph node involvement).
* Absence of metastatic disease at a distance (computerized tomography, diagnostic laparoscopy and peritoneal lavage).
* Age 18-75 years.
* Clinical functionality by the ECOG scale between 0 and 1.
* Preserved renal function (creatinine clearance greater than 50 mL / min).
* Signature of Informed Consent Form

Exclusion Criteria:

* Active neoplasm of another primary site other than non-melanoma skin carcinoma.
* Lesions of the esophagogastric transition
* Unresectable lesions by computed tomography and / or diagnostic laparoscopy.
* Obstructive tumors (acute intestinal occlusion or subocclusion).
* Tumors with signs of significant or persistent bleeding.
* Carcinoma in situ.
* Different histological type of adenocarcinoma.
* Gastric stump tumors.
* Previous chemotherapeutic or radiotherapy treatment.
* Current pregnancy or breastfeeding.
* Total bilirubin above 1.5mg / dL.
* Hepatic transaminases greater than 1.5 times the upper limit of normality.
* Decompensated and / or symptomatic cardiomyopathy: congestive heart failure with functional class greater than 2 by the New York Heart Association; active coronary disease; uncontrolled cardiac arrhythmia; history of acute myocardial infarction in the last 6 months.
* Psychological, familial, social or even geographical condition that potentially hinders adherence to the study protocol and the pre-established follow-up.
* Current or previous psychiatric or neurological diagnosis that is decompensated, compromises the cognition, functionality or adherence to the proposed treatment.
* Other comorbidities that are decompensated at the time of treatment.
* Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2017-02-23 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | 4-8 weeks after neoadjuvant chemotherapy complete
  To evaluate the Pathologic Complete Response (pCR).

SECONDARY OUTCOMES:
Disease-free survival (DFS) | At 2, 3 and 5 years after preoperative treatment with FOLFIRINOX regimen.
  Evaluate Disease-free survival (DFS).
Overall survival (OS) | At 2, 3 and 5 years after preoperative treatment with FOLFIRINOX regimen.
  Evaluate Overall survival (OS).
R0-resection rate | 4-8 weeks after neoadjuvant chemotherapy complete
  Evaluate the R0 resection rate (absence of microscopic residual disease).
Rate of Treatment Completion | 4-8 weeks after neoadjuvant chemotherapy complete
  Evaluate the rate of completion of treatment (chemotherapy and surgical approach).
Rate of adverse events | Through neoadjuvant chemotherapy (4 months)
  Rate and description of adverse events
Rate of Disease Progression | Through neoadjuvant chemotherapy (4 months)
  Evaluate the rate of disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided